CLINICAL TRIAL: NCT05282693
Title: Ergogenic Properties of Magnesium Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Bell (Other)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1659
Record Dates: First submitted 2022-01-26; First posted 2022-03-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Exercise Performance; Gut -Microbiota; Mitochondrial Function
MeSH Terms: interventions — Magnesium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either placebo for 9-days of the intervention separated by a 3-week washout period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Coded bottles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReMag (Experimental): Liquid Lemon flavor drink containing 300 mg magnesium chloride (Regmag) consumed twice daily for 9 days
  Interventions: Dietary Supplement: ReMag
- ReMag Placebo (Placebo Comparator): Liquid Lemon flavor drink placebo comparator consumed twice daily for 9 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ReMag — 300 mg of ReMag dissolved in lemon flavor liquid
  Other Names: Magnesium Chloride
  Arms: ReMag
Dietary Supplement: Placebo — Lemon flavored liquid
  Arms: ReMag Placebo

SUMMARY:
The purpose of the proposed project is to determine if short-term dietary supplementation of magnesium will improve performance during a series of lab-based exercise tests, will favorably modify the gut-microbiota, and will augment skeletal muscle mitochondrial function.

DETAILED DESCRIPTION:
Magnesium is the fourth most abundant mineral in the human body. It is critical to day-to-day physiological function including the regulation of metabolism, cardiovascular function, immune function, and the operation of the nervous system. In light of its important role in physiology, dietary supplementation of magnesium has been purported to improve athletic performance, although the precise mechanism is unclear. The foci of the proposed study is the ergogenic effects of magnesium, its potential influence on gut health, and its potential ability to improve skeletal muscle function. The investigators will be studying an athletic/competitive population of endurance-trained adults. This group is likely to be the most interested in the use of magnesium to enhance athletic performance. Also, by only recruiting habitual exercisers, the variability between participants is likely to be reduced compared with if the investigators had also recruited people who are usually sedentary.

ELIGIBILITY:
Inclusion Criteria:

* Competitive cyclists
* Adult males and females (18 - 40 years, inclusive) who have exercised a minimum of 5 days per week, for a minimum of 30-minutes/session, during the previous 2 years.
* Maximal oxygen uptake (VO2max) satisfying the minimum criteria for "Good" (sex- and age-adjusted) as defined by the American College of Sports Medicine.

Exclusion Criteria:

* Identification of a contra-indication to exercise during a 12-lead exercise stress test
* Use of a magnesium supplement within the previous 4 weeks
* Pregnancy or breast-feeding
* Unable to perform vigorous exercise
* History (previous diagnosis) of kidney disease
* Use of laxatives, Zinc, diuretics, proton pump inhibitors, over the counter agents such as certain heartburn and GI/gut treatments (laxatives) which contain magnesium, Zinc or other high dose cations which reduce absorption of Magnesium

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of completion of time trial to placebo | After 9 days of intervention
  Amount of time it takes to cycle 10 kilometers
Comparison of power output to placebo | After 9 days of intervention
  Cycling for 30 seconds
Comparison of indirect Calorimetry (VO2max) to placebo | After 8 days of intervention
  During a standard stress test VO2 max will be measured
Comparison of lactate threshold to placebo | After 8 days of intervention
  During a standard stress test lactate threshold will be measured
Comparison of Mitochondrial Function to placebo | After 8 days of intervention
  Assessed via high-resolution mitochondrial respirometry in permeabilized skeletal muscle.
Comparison of Shannon and Faith's microbiota diversity scores in feces to placebo | After 9 days of intervention,
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
Calculation and ordination of B-diversity scores for all fecal samples to assess clustering | After 9 days of intervention
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
Determination of differentially abundant microbiota in feces of collected during treatment compared to placebo | After 9 days of intervention
  Assessed via 16s ribosomal ribonucleic acid microbial profiling
Comparison of abundant microbiota to markers in feces to placebo | After 9 days of intervention
  Assessed via Linear discriminant analysis Effect Size algorithm
Comparison Human Granulocyte Macrophage Colony-Stimulating Factor to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interferon gamma to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 1 beta to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 2 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 4 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 5 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 6 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 7 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 8 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 10 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 12 (p70) to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison interleukin 13 to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison Tumor Necrosis Factor alpha to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel
Comparison High-sensitivity C-reactive protein to placebo | After 9 days of intervention
  Assessed via 13-plex human T-cell cytokine panel

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States